CLINICAL TRIAL: NCT00859807
Title: A Bioequivalence Study Comparing Camoquin® Suspension (Pfizer) To Flavoquine® Tablets (Sanofi Aventis) In Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B0731001
Record Dates: First submitted 2009-03-06; First posted 2009-03-11 (Estimated); Last update posted 2010-04-21 (Estimated); Status verified 2010-04

CONDITIONS: Falciparum Malaria
Keywords: Amodiaquine suspension; Flavoquine tablets; Bioequivalence study
MeSH Terms: conditions — Malaria, Falciparum | interventions — Amodiaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (19 subjects) (Experimental): Period 1: treatment A (15.3 mL (50 mg/5 mL) AQ suspension (Pfizer); test treatment.
  Period 2: treatment B (1 x 200 mg tablet Flavoquine® (Sanofi Aventis); reference treatment).
  Interventions: Drug: Flavoquine®, Camoquin® Suspension
- Sequence 2 (19 subjects) (Experimental): Period 1: treatment B (1 x 200 mg tablet Flavoquine® (Sanofi Aventis Period 2: treatment A (15.3 mL (50 mg/5 mL) AQ suspension (Pfizer); test treatment
  Interventions: Drug: Flavoquine®, Camoquin® Suspension

INTERVENTIONS:
Drug: Flavoquine®, Camoquin® Suspension — Treatment A 15.3 mL (50 mg/5 mL) AQ suspension single dose. Treatment B (1 x 200 mg tablet Flavoquine® (Sanofi Aventis) single dose.
  Other Names: amodiaquine
  Arms: Sequence 1 (19 subjects)
Drug: Flavoquine®, Camoquin® Suspension — Treatment A 15.3 mL (50 mg/5 mL) AQ suspension single dose. Treatment B (1 x 200 mg tablet Flavoquine® (Sanofi Aventis) single dose.
  Other Names: amodiaquine
  Arms: Sequence 2 (19 subjects)

SUMMARY:
The purpose of this study is to determine bioequivalence of amodiaquine suspension ( Pfizer) and the WHO approved reference product Flavoquine® tablet ( Sanofi Aventis).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive.
* Body Mass Index (BMI) of 18 to 30 kg/m2; and a total body weight >45 kg (99 lbs).
* An informed consent document signed and dated by the subject or a legally acceptable representative.

Exclusion Criteria:

* A history of drug induced agranulocytosis and history of liver and hematological problems while taking amodiaquine.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2009-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Cmax, AUCtlast and AUCinf for amodiaquine. | end of study

SECONDARY OUTCOMES:
Cmax and AUC72 for DesethylAQ | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Navi Mumbai, Maharashtra, India

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0731001&StudyName=A%20Bioequivalence%20Study%20Comparing%20Camoquin%AE%20Suspension%20%28Pfizer%29%20To%20Flavoquine%AE%20Tablets%20%28Sanofi%20Aventis%29%20In%20Healthy%20Subjects%0A%0A